CLINICAL TRIAL: NCT02408133
Title: Effectiveness of Home-based Exercise in Quality of Life and Physical Fitness in Older Woman in Breast Cancer Treatment: Randomized Clinical Trial
Brief Title: Effectiveness of Home-based Exercise in Quality of Life and Physical Fitness in Older Woman in Breast Cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, José Roberto da Silva Junior, Master in Health, Professor Fernando Figueira Integral Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1165-5043
Record Dates: First submitted 2015-02-24; First posted 2015-04-03 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; elderly; quality of life; exercise
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): The control group will be accompanied according to the service routine.
- Exercise (Experimental): The group will be instructed to perform home exercises autonomously for range of motion and muscular fitness
  Interventions: Other: Home exercise

INTERVENTIONS:
Other: Home exercise — Will be offered to the group, instructional material (manual exercises) and point you to an exercise routine to be performed independently for range of motion and muscular fitness, using the environmental resources of the same household. A daily frequency in performing this exercise routine is suggested. Also, be given incentives and guidelines for the practice of active commuting (walking) to be accumulated at least 10 to 20 minutes of this activity daily. All control guidelines and training for the use of the exercise manual will be offered through an introductory lecture and subsequent weekly telephone contacts (2 times a week). The participants in this group should fulfill their respective program for a total period of 12 weeks.
  Other Names: Exercise
  Arms: Exercise

SUMMARY:
The purpose of this study is to evaluate the effectiveness of home exercise on quality of life and physical fitness of elderly women with breast cancer patients undergoing cancer treatment.

DETAILED DESCRIPTION:
Cancer has excelled as a leading cause of mortality. It is particularly serious in the elderly due to increased risk of functional impairment and present comorbidities. The physical exercise appears as a promising intervention in the various stages of the treatment, mitigating the adverse effects in short- and long-term the oncologic treatment. Its regular practice after a diagnosis of breast cancer is associated with 40 % to 50 % lower rates of mortality. Produces metabolic and morphological changes that may make it an important option in the treatment, prevention, and recovery process of these patients. In this context the present study aims to verify the effectiveness of home exercise on quality of life and physical fitness of elderly undergoing treatment for breast cancer. This study it's a Randomized Clinical Trial. Data will be collected at the Department of Oncology at the Professor Fernando Figueira Integral Medicine Institute (IMIP), which serves patients in the public health system (SUS) from the metropolitan area of Recife, State of Pernambuco. will be held from March to December 2015. Will be studied elderly diagnosed with breast cancer undergoing treatment in the Adult Oncology Service of IMIP. For the analysis of means and frequencies, the investigators intend to use descriptive statistics and the results will be displayed in graphs and tables. For inferential statistical analysis, the investigators intend to use the Student's t test, or the Mann - Whitney test, according to the normality of the sample. For categorical variables, contingency tables are constructed of type 2x2. Chi-square tests of association with Yates correction and Fisher's exact test will be used. The risk ratio (RR) will be calculated as a measure of the relative risk of different outcomes according to the realization of one or another approach to exercise and control group. The Software Stata 12.0 will be used for data processing and will be accepted at p < 0,05. The project meets the requirements of the National Board of Health and was approved by the IMIP Research Ethics Committee. Patients who agree to sign the Instrument of Consent will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer diagnosis with stage I or II;
* Being in treatment for breast cancer (chemotherapy; radiotherapy and / or hormone therapy).

Exclusion Criteria:

* Absolute contraindication for physical exercises;
* Severe depression diagnosis using the Geriatric Depression Scale;
* Malnutrition (wasting grades I, II and III), detected by body mass index (BMI), according to the WHO criteria.

Ages: 60 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Variation in the performance of Lift and Sitting Test | Change from Baseline in Lift and Sitting Test and after 12 weeks
  Test which comprises the Battery Senior Fitness Test (SFT). Evaluates the Lower body strength according to the number of times the individual stood up and sat down in 30 seconds. Characterized as continuous numeric variable.
Variation in the performance of Flexion forearm Test | Change from Baseline in Flexion forearm Test and after 12 weeks
  Test which comprises the Battery Senior Fitness Test (SFT). Evaluates the upper body strength according to the number of push-ups of forearm in 30 seconds. Characterized as continuous numeric variable.
Variation in the performance of Six Minute Walk Test (6MWT) | Change from Baseline in Six Minute Walk Test (6MWT) and after 12 weeks
  Test which comprises the Battery Senior Fitness Test (SFT). Evaluates aerobic endurance. Total meters walked for 6 minutes walk. Characterized as continuous numeric variable.
Variation in the performance of March Stationary two minutes Test | Change from Baseline in March Stationary two minutes Test and after 12 weeks
  Test which comprises the Battery Senior Fitness Test (SFT). Evaluates aerobic endurance (alternative test). Total double past stationary in 2 minutes. Characterized as continuous numeric variable.
Variation in the performance of Skip and Vir 2.44 meters test | Change from Baseline in Skip and Vir 2.44 meters test and after 12 weeks
  Test which comprises the Battery Senior Fitness Test (SFT). Assesses motor agility and dynamic balance. Evaluates the time in seconds and hundredths in an established path of 2.44 meters on the route to go and return to starting position. Characterized as continuous numerical variable.
Variation in the performance of Sit and Reach Modified test (In the Chair) | Change from Baseline in Sit and Reach Modified test (In the Chair) and after 12 weeks
  Test which comprises the Battery Senior Fitness Test (SFT). Evaluates the lower hemisphere flexibility. distance in centimeters reached the tip of the middle fingers and the floor in the sitting position. Characterized as continuous numerical variable.
Variation in the performance of Flexibility test of the upper limbs | Change from Baseline in Flexibility test of the upper limbs and after 12 weeks
  Test which comprises the Battery Senior Fitness Test (SFT). Evaluates the flexibility of the upper limbs. It measures the distance in centimeters between the tips of the fingers in the back area. Characterized as continuous numeric variable.
Body Mass Index | Change from Baseline in Body Mass Index and after 12 weeks
  the calculation will be determined by the ratio between the weight (in kilograms) and the square of height (in meters). Characterized as continuous numeric variable
Variation in the performance of Muscle strength Test | Change from Baseline in Muscle strength Test after 12 weeks
  Hand Grip Strength Test. Continuous numeric variable: average kilogram-force (KgF)

SECONDARY OUTCOMES:
Quality of life | Change from Baseline in Quality of life after 12 weeks
  Numeric variable: average score from 0 to 100 for 30 issues of questionnaire developed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)

OTHER OUTCOMES:
Weight | Change from Baseline in Weight after 12 weeks
  Measurement of body mass, using electronic scale Tanita®. Characterized as continuous numerical variable, measured in kilograms
Height | Change from Baseline in Height after 12 weeks
  Greater distance between the vertex and the ground when the individual in the standing position, using the stadiometer Sanny® brand. Characterized as continuous numeric variable measured in meters
Total Muscle Mass Index (IMMT) | Change from Baseline in Total Muscle Mass Index (IMMT) after 12 weeks
  Measure of muscle mass relative amount contained in the body, through perimetry using anthropometric tape Sanny® brand. Characterized as continuous numeric variable.
Fat percentage | Change from Baseline in Fat percentage after 12 weeks
  as the relative amount of fat contained in the body by means of perimetry using anthropometric Sanny® tape mark. Characterized as continuous numeric variable.

CONTACTS AND LOCATIONS:
Overall Officials: João Guilherme Bezerra Alves, Doctor, Study Director — Instituto de Medicina Integral Prof. Fernando Figueira; Breno Augusto Bormann de Souza Filho, Graduate, Principal Investigator — Instituto de Medicina Integral Prof. Fernando Figueira; José Roberto da Silva Junior, Master, Study Director — Instituto de Medicina Integral Prof. Fernando Figueira; William Serrano Smethurst, Master, Study Director — Instituto de Medicina Integral Prof. Fernando Figueira; JuremaTelles de Oliveira Lima, Master, Study Director — Instituto de Medicina Integral Prof. Fernando Figueira